CLINICAL TRIAL: NCT04957927
Title: Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Usama Azhar (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Sponsor-Investigator, Usama Azhar, Post Graduate Resident in Pediatrics(MD Pediatrics), King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 747/RC/KEMU
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis in children; Montelukast; Intranasal Fluticasone Propionate
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Fluticasone Propionate Group (Experimental): Intranasal Fluticasone Propionate 50mcg/actuation in each nostril 24 hourly
  Interventions: Drug: Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age
- Montelukast Group (Experimental): Montelukast 4mg oral granule formulation 24 hourly
  Interventions: Drug: Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age

INTERVENTIONS:
Drug: Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age — Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age

SUMMARY:
To determine the Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age.

DETAILED DESCRIPTION:
Our study will compare the Effectiveness of Montelukast Versus Intranasal Fluticasone Propionate in the Management of Allergic Rhinitis Among Children 02 to 05 Years of Age as in our population compliance with oral medication is better among patients, and is socially and culturally more acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Age:02 to 05 Years of Age
* both genders will be included.
* patients diagnosed with allergic rhinitis.

Exclusion Criteria:

* patients older than 05 years of age
* a positive history of HIV,TB,Immune deficiency.
* any nasal structural abnormality i.e.polyps,deviated nasal septum.
* history of frequent nasal bleeding,epistaxis.
* concomitant asthma.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-09-12 (Estimated); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Day and Night time nasal symptoms score of Allergic Rhinitis | 2 months
  Effectiveness will be assessed by noticing the Improvement in Day and Night time nasal symptoms score of Allergic Rhinitis.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Haroon Hamid, MBBS,FCPS,FRCS, Principal Investigator — Chairman/Head of Department of pediatrics unit 1 K.E. Medical University/Mayo hospital lahore
Locations (1):
- King Edward Medical University/Mayo hospital lahore,punjab,pakistan 54000, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Emeryk A, Emeryk-Maksymiuk J, Janeczek K. New guidelines for the treatment of seasonal allergic rhinitis. Postepy Dermatol Alergol. 2019 Jun;36(3):255-260. doi: 10.5114/ada.2018.75749. Epub 2019 Jun 18. PMID 31333340
- [Background] Chong SN, Chew FT. Epidemiology of allergic rhinitis and associated risk factors in Asia. World Allergy Organ J. 2018 Aug 6;11(1):17. doi: 10.1186/s40413-018-0198-z. eCollection 2018. PMID 30128063
- [Background] Al-Digheari A, Mahboub B, Tarraf H, Yucel T, Annesi-Maesano I, Doble A, Lahlou A, Tariq L, Aziz F, El Hasnaoui A. The clinical burden of allergic rhinitis in five Middle Eastern countries: results of the SNAPSHOT program. Allergy Asthma Clin Immunol. 2018 Nov 19;14:63. doi: 10.1186/s13223-018-0298-x. eCollection 2018. PMID 30473712
- [Background] May JR, Dolen WK. Management of Allergic Rhinitis: A Review for the Community Pharmacist. Clin Ther. 2017 Dec;39(12):2410-2419. doi: 10.1016/j.clinthera.2017.10.006. Epub 2017 Oct 25. PMID 29079387
- [Background] Jindal A, Suriyan S, Sagadevan S, Narasimhan M, Shanmuganathan A, Vallabhaneni V, Rajalingam R. Comparison of Oral Montelukast and Intranasal Fluticasone in Patients with Asthma and Allergic Rhinitis. J Clin Diagn Res. 2016 Aug;10(8):OC06-10. doi: 10.7860/JCDR/2016/20741.8268. Epub 2016 Aug 1. PMID 27656477
- [Background] Seidman MD, Gurgel RK, Lin SY, Schwartz SR, Baroody FM, Bonner JR, Dawson DE, Dykewicz MS, Hackell JM, Han JK, Ishman SL, Krouse HJ, Malekzadeh S, Mims JW, Omole FS, Reddy WD, Wallace DV, Walsh SA, Warren BE, Wilson MN, Nnacheta LC; Guideline Otolaryngology Development Group. AAO-HNSF. Clinical practice guideline: Allergic rhinitis. Otolaryngol Head Neck Surg. 2015 Feb;152(1 Suppl):S1-43. doi: 10.1177/0194599814561600. PMID 25644617
- [Background] Goh BS, Ismail MI, Husain S. Quality of life assessment in patients with moderate to severe allergic rhinitis treated with montelukast and/or intranasal steroids: a randomised, double-blind, placebo-controlled study. J Laryngol Otol. 2014 Mar;128(3):242-8. doi: 10.1017/S002221511400036X. Epub 2014 Mar 11. PMID 24618303
- [Background] Mansi N, D'Agostino G, Scire AS, Morpurgo G, Gregori D, Gulati A, Damiani V. Allergic Rhinitis in Children: A Randomized Clinical Trial Targeted at Symptoms. Indian J Otolaryngol Head Neck Surg. 2014 Dec;66(4):386-93. doi: 10.1007/s12070-014-0708-4. Epub 2014 Feb 11. PMID 26396949
- [Background] Roberts G, Xatzipsalti M, Borrego LM, Custovic A, Halken S, Hellings PW, Papadopoulos NG, Rotiroti G, Scadding G, Timmermans F, Valovirta E. Paediatric rhinitis: position paper of the European Academy of Allergy and Clinical Immunology. Allergy. 2013 Sep;68(9):1102-16. doi: 10.1111/all.12235. Epub 2013 Aug 19. PMID 23952296
- [Background] Ologe FE, Adebola SO, Dunmade AD, Adeniji KA, Oyejola BA. Symptom score for allergic rhinitis. Otolaryngol Head Neck Surg. 2013 Apr;148(4):557-63. doi: 10.1177/0194599813477605. Epub 2013 Feb 21. PMID 23429039
- [Background] Herr M, Clarisse B, Nikasinovic L, Foucault C, Le Marec AM, Giordanella JP, Just J, Momas I. Does allergic rhinitis exist in infancy? Findings from the PARIS birth cohort. Allergy. 2011 Feb;66(2):214-21. doi: 10.1111/j.1398-9995.2010.02467.x. Epub 2010 Aug 30. PMID 20804465
- [Background] Hardjojo A, Shek LP, van Bever HP, Lee BW. Rhinitis in children less than 6 years of age: current knowledge and challenges. Asia Pac Allergy. 2011 Oct;1(3):115-22. doi: 10.5415/apallergy.2011.1.3.115. Epub 2011 Oct 11. PMID 22053307
- [Background] Phan H, Moeller ML, Nahata MC. Treatment of allergic rhinitis in infants and children: efficacy and safety of second-generation antihistamines and the leukotriene receptor antagonist montelukast. Drugs. 2009;69(18):2541-76. doi: 10.2165/9884960-000000000-00000. PMID 19943707
- [Background] Ratner PH, Howland WC 3rd, Arastu R, Philpot EE, Klein KC, Baidoo CA, Faris MA, Rickard KA. Fluticasone propionate aqueous nasal spray provided significantly greater improvement in daytime and nighttime nasal symptoms of seasonal allergic rhinitis compared with montelukast. Ann Allergy Asthma Immunol. 2003 May;90(5):536-42. doi: 10.1016/S1081-1206(10)61847-9. PMID 12775135
- [Background] Nayak AS, Philip G, Lu S, Malice MP, Reiss TF; Montelukast Fall Rhinitis Investigator Group. Efficacy and tolerability of montelukast alone or in combination with loratadine in seasonal allergic rhinitis: a multicenter, randomized, double-blind, placebo-controlled trial performed in the fall. Ann Allergy Asthma Immunol. 2002 Jun;88(6):592-600. doi: 10.1016/S1081-1206(10)61891-1. PMID 12086367